CLINICAL TRIAL: NCT05008081
Title: An International Multi-centre Prospective Cohort Study in Patients Hospitalized for an Acute Exacerbation of COPD
Brief Title: The CATALINA Study
Status: Recruiting | Type: Observational
Sponsor: Wim Janssens (Other)
Collaborators: European Respiratory Society (Other); AstraZeneca (Industry); Roche Pharma AG (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Wim Janssens, MD, PhD, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S64324
Record Dates: First submitted 2021-08-06; First posted 2021-08-17 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation
Keywords: COPD; Exacerbation; Hospitalization
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — * Blood (serum/plasma)
  * Sputum
  * Nasopharygeal swab
  * Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CATALINA study is a prospective cohort study embedded within CICERO (Collaboration In COPD ExaceRbatiOns, a European Respiratory Society supported Clinical Research Collaboration), designed to collect standardised, longitudinal clinical data and biological samples in 20 centres across Europe and beyond.

DETAILED DESCRIPTION:
The initial objective is to recruit 1000 patients hospitalised for an acute COPD exacerbation by the end of CICERO's first lifecycle (3 years), from whom 1 year follow-up data and biological samples will be collected. By doing so, CICERO aims to develop a comprehensive European COPD patient data- and biobank phenotyped in relation to the exacerbation, to support the development of future EU-wide clinical intervention trials in COPD for specific patient subgroups, as well as new prognostication tools for COPD exacerbations.

The clinical data and biological samples will be obtained during 6 scheduled study visits, during the hospitalization period of the index acute exacerbation as well as the outpatient setting after hospital discharge; and 3 additional unscheduled study visits should the patient be readmitted for respiratory reasons during study participation (i.e. first readmission only).

* 3 study visits will be scheduled during the hospitalization period of the index acute exacerbation:

  * visit 1: within 48h of hospital admission, study inclusion (Day 1)
  * visit 2: at 72h after study inclusion (Day 3)
  * visit 3: at hospital discharge, at investigator's discretion (Day X)
* 3 study visits will be scheduled during the outpatient setting:

  * visit 4: at 3 months after study inclusion (Day 90)
  * visit 5: at 6 months after study inclusion (Day 180)
  * visit 6: at 12 months after study inclusion (Day 365)
* The first hospital readmission for respiratory reasons during the patient's study participation will undergo the same testing schedule as mandated during the hospitalization period of the index event:

  * unscheduled visit 1: within 48h of first hospital readmission
  * unscheduled visit 2: within 72h of first hospital readmission
  * unscheduled visit 3: at hospital discharge for first hospital readmission

Resulting from CICERO's future lifecycles will be the continued expansion of the data- and bio-bank, both in cohort size and duration of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Established diagnosis of COPD by medical doctor (based on clinical history OR pulmonary function test with an FEV1/FVC < 0.7)
* Current hospitalization with suspicion of an acute exacerbation of COPD (AECOPD)
* Inclusion within 48 hours post hospital admission
* Voluntary written informed consent of the participant or his/her representative obtained prior to any study procedure

Exclusion Criteria:

* Patients unwilling or unable to comply with study procedures
* Patients not requiring treatment with systemic corticosteroids, antibiotics or both as a minimum therapy for the index AECOPD
* Patients with a confirmed positive test result for COVID19, or those highly suspected based on clinical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD, hospitalized for an acute exacerbation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Will be assessed during 1 year, on visits 2-6
  Death from any cause

SECONDARY OUTCOMES:
Step-up in hospital care for respiratory reasons | Will be assessed during 1 year, on visits 2-6
  A composite outcome measure defined as:
  1. New hospitalization for respiratory reasons
  2. Hospital care intensification from baseline (ie. within 24h from hospital admission) for respiratory reasons, including:
     * 2.1 Non-invasive respiratory therapy (oxygen by mask or nasal flow)
     * 2.2 Non-invasive respiratory therapy (oxygen by NIV or high flow)
     * 2.3 Invasive respiratory therapy (intubation and mechanical ventilation)
     * 2.4 Physiological support with inotropes
Treatment intensification for respiratory reasons | Will be assessed during 1 year, on visits 2-6
  A composite outcome measure defined as:
  1. Prolongation of systemic corticosteroids >5 days administered for the index acute exacerbation or first readmission for respiratory reasons
  2. Upgrade of antibiotics administered for the index exacerbation or first readmission for respiratory reasons
  3. New course of systemic corticosteroids for respiratory reasons
  4. New course of antibiotics for respiratory reasons
Treatment failure | Will be assessed during 1 year, on visits 2-6
  A composite outcome measure defined as:
  1. All-cause mortality
  2. Step-up in hospital care for respiratory reasons
  3. Treatment intensification for respiratory reasons
Severe treatment failure | Will be assessed during 1 year, on visits 2-6
  As intensification of drug treatment regimens and treatment intensifications are country/region-specific and not always related to failure of disease control, severe treatment failure (STF) will be defined as the composite of:
  1. All-cause mortality
  2. Step-up in hospital care for respiratory reasons
Readmission for a severe COPD exacerbation | Will be assessed during 1 year, on visits 2-6
  Readmission of the patient to the hospital for a severe COPD exacerbation
New hospitalization for respiratory reasons | Will be assessed during 1 year, on visits 2-6
  New admission of the patient to the hospital for respiratory reasons
Hospital care intensification for respiratory reasons | Will be assessed during 1 year, on visits 2-6
  A composite outcome measure defined as:
  1. Non-invasive respiratory therapy (oxygen by mask or nasal flow)
  2. Non-invasive respiratory therapy (oxygen by NIV or high flow)
  3. Invasive respiratory therapy (intubation and mechanical ventilation)
  4. Physiological support with inotropes
Time to | Will be assessed during 1 year, on visits 2-6
  The time to the following outcomes will be measured:
  1. All-cause mortality
  2. First hospital readmission for respiratory reasons
  3. Hospital care intensification for respiratory reasons
  4. Treatment intensification for respiratory reasons
  5. Treatment failure
  6. Severe treatment failure
Number of participants with a new or changed Do Not Resuscitate (DNR) code | Will be assessed during 1 year, on visits 2-6
  The implementation of a new or changed DNR code during study participation will be measured.
  * DNR 0: do not restrict therapy (i.e. explicit statement not to withhold any life-sustaining interventions)
  * DNR 1: do not resuscitate, further specified as:
  DNR 1a: No CPR DNR 1b: No CPR + no intubation + NIV to be considered
  * DNR 2: do not extend therapy (i.e. no CPR + no intubation + no NIV)
  * DNR 3: discontinue therapy (i.e. no CPR + no intubation + no NIV + withdrawal of current treatment°)
  Abbreviations: CPR, cardiopulmonary resuscitation; NIV, non-invasive ventilation; °, treatment of disabling symptoms to be prioritised, however, no life-prolonging interventions are to be continued
Cumulative dose of systemic corticosteroids | Will be assessed during 1 year, on visits 2-6
  The total dose of systemic corticosteroids administered during study participation will be measured.
Total days in hospital | Will be assessed during 1 year, on visits 2-6
  Total number of days spent in a hospital during study participation will be measured.
Change in modified Medical Research Council (mMRC): a dyspnea scale | Will be assessed during 1 year, on visits 2-6
  The change in the following patient reported outcome measures (PROM) will be measured:
  modified Medical Research Council (mMRC): a dyspnea scale
  * scale: 0 to 4
  * interpretation: higher scores indicate worse outcome
Change in COPD Assessment Test (CAT): a COPD impact scale | Will be assessed during 1 year, on visits 2-6
  The change in the following patient reported outcome measures (PROM) will be measured:
  COPD Assessment Test (CAT): a COPD impact scale
  * scale: 0 to 40
  * interpretation: higher scores indicate worse outcome
Change in Patient Health Questionnaire-9 (PHQ-9): a depression scale | Will be assessed during 1 year, on visits 2-6
  The change in the following patient reported outcome measures (PROM) will be measured:
  Patient Health Questionnaire-9 (PHQ-9): a depression scale
  * scale: 0 to 29
  * interpretation: higher scores indicate worse outcome
Change in Generalized Anxiety Disorder-7 (GAD-7): an anxiety scale | Will be assessed during 1 year, on visits 2-6
  The change in the following patient reported outcome measures (PROM) will be measured:
  Generalized Anxiety Disorder-7 (GAD-7): a anxiety scale
  * scale: 0 to 21
  * interpretation: higher scores indicate worse outcome
Change in patient reported experience measure (PREM) | Will be assessed during 1 year, on visits 2-6
  The change in the following PREM will be measured:
  1. Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS): measuring patients' perceptions of their hospital experience
  -interpretation: higher scores indicate better outcome
Change in comorbidities | Will be assessed during 1 year, on visits 2-6
  Changes in baseline comorbidies (ie. the appearance of new or worsening of existing) will be measured
Change in biomarker Eotaxin-3 (CCL26) | Will be assessed during 1 year, on visits 2-6
  Eotaxin-3 is a small cytokine belonging to the CC chemokine family (called CCL26, Chemokine (C-C motif) ligand 26). Eotaxin-3 is chemotactic for eosinophils and basophils and elicits its effects by binding to the cell surface chemokine receptor CCR3.
Change in biomarker IL-5 | Will be assessed during 1 year, on visits 2-6
  Interleukin-5 (IL-5) acts on mature eosinophils, leading to proliferation, activation, differentiation, and survival; playing a critical role in the host immune response to infections.
Change in biomarker IL-33 | Will be assessed during 1 year, on visits 2-6
  Interleukin-33 (IL-33) is described as an inducer of type 2 immune responses, activating T helper 2 cells and mast cells.
Change in biomarker MCP-4 (CCL13) | Will be assessed during 1 year, on visits 2-6
  Monocyte chemotactic protein 4 (MCP-4), also called CCL13, is a major chemo-attractant for eosinophils, basophils, monocytes and T lymphocytes
Change in biomarker TARC4 (CCL17) | Will be assessed during 1 year, on visits 2-6
  Thymus and activation regulated chemokine (TARC), also known as CCL17, is a chemokine that induces chemotaxis of Type 2 T helper (Th2) cells.
Change in biomarker IP-10 (CXCL10) | Will be assessed during 1 year, on visits 2-6
  Interferon gamma-induced protein 10 (IP-10 (CXCL10)) chemoattracts Th1 lymphocytes and monocytes, and inhibits cytokine-stimulated hematopoietic progenitor cell proliferation.
Change in biomarker IL1A | Will be assessed during 1 year, on visits 2-6
  Interleukin 1 alpha (IL1A) stimulates the activity of genes involved in inflammation and immunity
Change in biomarker IL-8 | Will be assessed during 1 year, on visits 2-6
  Interleukin 8 (IL-8) is a chemokine produced by macrophages and other cell types such as epithelial cells, airway smooth muscle cells and endothelial cells; which attracts and activates neutrophils in inflammatory regions
Change in biomarker GM-CSF | Will be assessed during 1 year, on visits 2-6
  Granulocyte-macrophage colony-stimulating factor (GM-CSF) regulates proliferation and/or activation of monocytes, macrophages, neutrophils and eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD, PhD, Study Chair — UZ/KU Leuven - Belgium; Mona Bafadhel, MD, PhD, Study Chair — King's College London - UK
Locations (18):
- Kepler University Hospital, Linz, Austria
- Belgium (3):
  - CHU St-Pierre Brussels, Brussels
  - UZ Leuven, Leuven
  - CHU UCL Namur Site Godinne, Yvoir
- France (2):
  - CHU de Lille, Lille
  - Cochin Hospital, Paris
- Germany (3):
  - LungenClinic, Großhansdorf
  - Klinikum Itzehoe, Itzehoe
  - University Medical Centre of Gießen & Marburg, Marburg
- University Hospital of Ferrara, Ferrara, Italy
- Netherlands (2):
  - UMC Groningen, Groningen
  - Maastricht University Medical Hospital, Maastricht
- Hospital Clinic de Barcelona, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (4):
  - Glenfield Hospital, Leicester
  - Guy's Saint Thomas, London
  - Royal Brompton Hospital, London
  - Churchil Hospital, Oxford

REFERENCES:
- See also: ERJ Editorial 2020 - The CICERO (Collaboration In COPD ExaceRbatiOns) Clinical Research Collaboration — https://pubmed.ncbi.nlm.nih.gov/32139591/
- See also: Int J COPD 2021 - Standardisation of Clinical Assessment, Management and Follow-Up of Acute Hospitalised Exacerbation of COPD: A Europe-Wide Consensus — https://pubmed.ncbi.nlm.nih.gov/33623379/
- See also: ERJ Open Research 2023 - Patients' Acceptance of Outcome and Experience Measurements During Hospitalisation for COPD Exacerbations: A Cicero CRC - ELF Online Patient Survey — https://openres.ersjournals.com/content/9/4/00148-2023
- See also: The CICERO website — https://www.cicero-copd.net/
- See also: The ERS - CICERO CRC webpage — https://www.ersnet.org/research/cicero---collaboration-in-copd-exacerbations